CLINICAL TRIAL: NCT00681746
Title: An Open Label Positron Emission Tomography (PET) Study With (11C)Flumazenil to Determine Central GABAA Receptor Occupancy of AZD6280 After Oral Administration to Healthy Volunteers
Brief Title: Positron Emission Tomography (PET) Study With (11C) Flumazenil to Determine Central GABAA Receptor Occupancy of AZD6280
Acronym: PET
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Mark A. Smith, MD, Medical Science Director, Emerging Psychiatry, AstraZeneca Pharmaceuticals
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: D0850C00011; EudractCT 2007-006683-29
Record Dates: First submitted 2008-05-16; First posted 2008-05-21 (Estimated); Last update posted 2010-12-10 (Estimated); Status verified 2008-11

CONDITIONS: Anxiety
Keywords: Anxiety; GABA receptors; Positron Emission Tomography; PET; phase I
MeSH Terms: conditions — Anxiety Disorders | interventions — 4-amino-8-(2,5-dimethoxyphenyl)-N-propylcinnoline-3-carboxamide; Flumazenil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: AZD6280; Drug: (11C) flumazenil

INTERVENTIONS:
Drug: AZD6280 — Single dose of oral solution or capsule(s). 3 times for the 2 subjects in Panel 1. Once for the 6 remaining subjects.
Drug: (11C) flumazenil — Single dose of intravenous solution. 4 times for 2 subjects in Panel 1. 2 times for the remaining 6 subjects. (once together with AZD6280)

SUMMARY:
The study is carried out in order to determine the relationship between the dose of AZD6280 and the blood concentration of AZD6280, and to investigate to which extent AZD6280 binds to GABAA receptors

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI) of 18-30 kg/m2 and weight of 60-100 kg
* Clinically normal physical findings, medical history and laboratory values.

Exclusion Criteria:

* Clinically significant illness or clinical relevant trauma within 2 weeks before the study start.
* History of clinically significant heart arrythmias or heart disease/problems.
* Previous participation in a PET study within the past 12 months. Suffer from claustrophobia and would be unable to undergo MRI (magnetic resonance imaging) or PET scanning.

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Estimated)
Dates: Start 2008-02; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Positron emission tomography using the radioligand (11C) flumazenil | 4 times per subject

SECONDARY OUTCOMES:
To assess safety of AZD7325 by assessment of adverse events, vital signs, ECGs, psychometric tests and laboratory variables. | 6 visits with tests for the 2 subjects in the first group (Panel 1). 4 visits with tests for the 6 remaining subjects. Some tests will be done several times per visit. All tests will not be done at every visit.
Investigate the pharmacokinetics of AZD6280 following single doses of AZD6280 by assessment of drug concentration in plasma. | 3 times for the 2 subjects in the first group (Panel 1). Once for the 6 remaining subjects. Up to 48 hours at each time.

CONTACTS AND LOCATIONS:
Overall Officials: Bo Fransson, Principal Investigator — AstraZeneca Clinical Pharmacology Unit, Stockholm, Sweden; Eva Taavo, Study Director — AstraZeneca R&D, Study Delivery, Clinical Development, Södertälje, Sweden
Locations (1):
- Research Site, Stockholm, Sweden

REFERENCES:
- [Derived] Jucaite A, Cselenyi Z, Lappalainen J, McCarthy DJ, Lee CM, Nyberg S, Varnas K, Stenkrona P, Halldin C, Cross A, Farde L. GABAA receptor occupancy by subtype selective GABAAalpha2,3 modulators: PET studies in humans. Psychopharmacology (Berl). 2017 Feb;234(4):707-716. doi: 10.1007/s00213-016-4506-4. Epub 2016 Dec 24. PMID 28013354